CLINICAL TRIAL: NCT04010487
Title: A Multi-omics Study on the Pathogenesis of Malignant Transformation of Adenomyosis
Brief Title: Multi-omics Study on the Pathogenesis of Malignant Transformation of Adenomyosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: AM-OMICS2
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Adenomyosis; Endometrial Cancer; Ectopic Endometrial Tissue; Eutopic Endometrium; Genomics; Transcriptomics
MeSH Terms: conditions — Adenomyosis; Endometrial Neoplasms | interventions — Exome Sequencing; Base Sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — This study acquired the formalin fixed paraffin-embedded (FFPE) tissue of patients pathologically conformed endometrial carcinoma arising in adenomyosis (EC-AIA) treated at Peking Union Medical College Hospital from July 15, 2017 to July 15, 2019. The formalin fixed paraffin-embedded tissues from patients pathologically diagnosed with adenomyosis during this time period were also included as control specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometrial carcinoma arising in adenomyosis: Patients pathologically conformed endometrial carcinoma arising in adenomyosis (EC-AIA)
  Interventions: Genetic: whole exome sequencing and RNA-sequencing
- Adenomyosis without malignancy: Patients pathologically diagnosed with adenomyosis
  Interventions: Genetic: whole exome sequencing and RNA-sequencing

INTERVENTIONS:
Genetic: whole exome sequencing and RNA-sequencing — The specimens from adenomyosis, endometrial cancer, and eutopic endometrium will be tested by whole exome sequencing and RNA-sequencing

SUMMARY:
This study is to explore the driving genes and the molecular mechanism of malignant transformation of adenomyosis. This study acquired the formalin fixed paraffin-embedded (FFPE) tissue of patients pathologically conformed endometrial carcinoma arising in adenomyosis (EC-AIA) treated at Peking Union Medical College Hospital from July 15, 2017 to July 15, 2019. The formalin fixed paraffin-embedded tissues from patients pathologically diagnosed with adenomyosis during this time period were also included as control specimens. The eutopic endometrium, normal adenomyosis tissue, and EC-AIA tissue were harvested from the FFPE tissue from patients with EC-AIA. The normal eutopic endometrium and normal adenomyosis tissue were obtained by laser microdissection. The driving genes and potential molecular mechanism of EC-AIA will be found by the technology of whole exome sequencing and transcriptomics (RNA-sequencing).

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed diagnosis with atypical hyperplasia and malignant transformation of adenomyosis glandular epithelium (including endometrioid, serous and clear cell carcinoma), with or without concurrent endometrial carcinoma
* Signed an approved informed consents

Exclusion Criteria:

* Not meeting all the inclusion criteria.
* The formalin fixed paraffin-embedded (FFPE) tissue was not acquired at the required time period.
* The patients enrolled had accompanied some other kinds of carcinoma (such as ovarian cancer, cervical cancer, primary peritoneal cancer).
* Patients had cancer history of certain organ (such as colorectal cancer, gastric cancer, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes two groups patients (about 22 cases in each group):
  * Patients pathologically conformed endometrial carcinoma arising in adenomyosis (EC-AIA)
  * Patients pathologically diagnosed with adenomyosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Frequencies of somatic driving mutations | One year
  The differences of distributions and frequencies of somatic driving mutations will be compared between eutopic ectopic endometrium, and cancer tissues by whole exome sequencing
Frequencies of alteration of RNA expression | One year
  The alteration of RNA expression, including mRNA, miRNA, and lncRNA will be compared between eutopic and ectopic endometrium, and cancer tissues by transcriptome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided